CLINICAL TRIAL: NCT02268734
Title: Molecular Profile of Metastatic Sporadic Medullary Thyroid Cancer (sMTC) Patients and Possible Correlation With Vandetanib Therapy
Brief Title: Molecular Profile of Metastatic Sporadic Medullary Thyroid Cancer Patients and Correlation With Vandetanib
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 178/13
Record Dates: First submitted 2014-09-04; First posted 2014-10-20 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Sporadic Medullary Thyroid Cancer
Keywords: Sporadic Medullary Thyroid Cancer Vandetanib miRNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — primary tumor and metastases tissue samples and other biological materials, including blood are collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sporadic Medullary Thyroid Cancer: Patients with diagnosis of locally relapsed and or metastatic sporadic MTC surgically treated (total thyroidectomy)

SUMMARY:
Vandetanib has been approved for patients with unresectable and/or metastatic medullary thyroid cancer (MTC) by the Food and Drug Administration, by the European Medicines Agency and, very recently, it has been licensed also by the Italian Regulatory Agency (AIFA) for the use in Italy. Vandetanib is an orally tyrosine kinase inhibitor (TKI) of vascular endothelial growth factor receptor (VEGFR), epidermal growth factor receptor (EGFR), and RET signaling.

Circulating microRNAs levels could be influenced by the treatment procedures and we hypothesize that a TKI therapy could influence the levels of circulating miRNAs as well.

Aim of this project is to seek non-invasive molecular markers potentially useful as prognostic tools for metastatic MTC patients.

DETAILED DESCRIPTION:
Medullary thyroid cancer (MTC) is considered worldwide a rare cancer. It derives from the parafolicular C-cells representing about 5-10% of all thyroid cancer. MTC is diagnosed as sporadic form (sMTC) in most of the patients, although in 20-30% of cases it could be hereditary and transmitted as an autosomal-dominant trait due to the germline mutations of the RET proto-oncogene. RET tyrosine kinase receptor is involved in the regulation of differentiation, proliferation, survival and cell motility processes through several intracellular signalling pathways, including MAPK and PI3K/AKT/mTOR pathways.

Vandetanib has been approved for patients with unresectable and/or metastatic MTC by the Food and Drug Administration, by the European Medicines Agency and, very recently, it has been licensed also by the Italian Regulatory Agency (AIFA) for the use in Italy. Vandetanib is an orally tyrosine kinase inhibitor (TKI) of vascular endothelial growth factor receptor (VEGFR), epidermal growth factor receptor (EGFR), and RET signaling. In a randomized phase III trial, response rate to vandetanib ranged from 31% to 55% with a predicted median progression-free survival (PFS) of 30.5 months while data on overall survival were still not available at the time of publication. These results suggest that approximately half of the patients could benefit from this compound whose activity is in every case limited in the time. Activity of vandetanib seems to be influenced by several factors, including RET mutational status and tumor genetic heterogeneity (clonal versus non-clonal RET mutation distribution). Recent analyses of circulating miRNAs in tumor patients have suggested that miRNA signatures may be useful as diagnostic/prognostic/predictive as well as pharmacodynamic markers for several tumor types.

No clinical neither biological data are currently available to identify which patients could really get a benefit from a TKI. In other words, some metastatic patients could suffer from an indolent disease, not requiring a TKI upfront and up to date, we are still not able to identify this selected group of patients Circulating miRNAs levels could be influenced by the treatment procedures, as it has been described in lung cancer where miR-21 and miR-24 resulted significantly lower in the post-operative period respect to the pre-operative one in paired samples. We hypothesize that a TKI therapy could influence the levels of circulating miRNAs as well.

Aim of this project is to seek non-invasive molecular markers potentially useful as prognostic tools for metastatic MTC patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of sMTC surgically treated (total thyroidectomy)
* locally relapsed and or metastatic sMTC
* metastatic MTC never treated with TKI before (valid for subjects treated with vandetanib only, in whom we will investigate the variation of circulating miRNA profile before and after vandetanib administration).

Exclusion Criteria:

* Patients with severe infection, active clinical co-morbidities, or a history of any other malignancy have been excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Petient with a diagnosis of sporadic locally relapsed and or metastatic medullary thyroid cancer surgically treated (total thyroidectomy) who adheres to a voluntary program of donation of own biological materials to a biorepository
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Validation of a miRNA profile | 8 months
  To validate the miRNA profile proposed by previous studies in sMTC in our series of metastatic sMTC
Define any correlations between the miRNA profiles and RET, and H- and K-RAS mutations | 8 months
  To assess whether there is any correlation between the miRNA profiles and RET, and H- and K-RAS mutations displayed by the same tumors
Define a circulating miRNA profile | 8 months
  To define a circulating miRNA profile in our series of metastatic sMTC and to assess whether miRNAs over-expressed in tumors are also present in plasma samples of the same sMTC patients
Analyze any change in circulating miRNAs | 8 months
  To analyze any change in circulating miRNAs profile according to the TKI treatment (vandetanib)
Correlate circulating miRNA profile with the burden of disease | 8 months
  To correlate circulating miRNA profile with the burden of disease and, possibly, with the genetic lesion of the primary tumors (RET and RAS mutations)
Evaluate the correlation between the response to vandetanib and the patients molecular profile | 8 months
  To evaluate the correlation between the response to vandetanib and the patients molecular profile including tissue miRNA, circulating miRNA and genetic lesion

CONTACTS AND LOCATIONS:
Overall Officials: Laura Locati, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Milan, Italy